CLINICAL TRIAL: NCT01267825
Title: A Randomized Trial of CT-guided Perineural Injection With a Corticosteroid Plus a Long Acting Local Anesthetic Versus Standard Medical Management in Patients With Acute Lumbar Radiculopathy and a Corresponding Disc Herniation
Brief Title: CT Guided Injection for Low Back Radiculopathy: A Randomized Clinical Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated early due to low enrollment. No data collected.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Prof. Emergency Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-06-162
Record Dates: First submitted 2010-10-25; First posted 2010-12-29 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Disc Herniation; Lumbosacral Radiculopathy
Keywords: Disc herniation; Lumbosacral radiculopathy; Corticosteroids
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT-guided intervention (Experimental): CT guided perineural injection of corticosteroid+ bupivicaine Also get typical medical care
  Interventions: Drug: CT-guided corticosteroid+ bupivicaine
- Standard medical care (Active Comparator)
  Interventions: Drug: Standard medical care

INTERVENTIONS:
Drug: CT-guided corticosteroid+ bupivicaine — CT-guided corticosteroid+ bupivicaine Also get standard medical care
  Arms: CT-guided intervention
Drug: Standard medical care — Naproxen + Oxycodone/ Acetaminophen
  Arms: Standard medical care

SUMMARY:
Herniated disc sometimes cause back pain radiating down to a leg. This pain can be so severe that it is functionally disabling. The purpose of this randomized clinical trial is to determine if corticosteroid medication, delivered directly to the area near the herniated disc, can improve the pain and functional disability associated with a herniated disc.

ELIGIBILITY:
Inclusion Criteria:

* Adults <60y
* < 1m of symptoms
* Symptoms consistent with herniated disc
* MRI demonstrates corresponding disc
* Back pain resulting in functional disability

Exclusion Criteria:

* Chronic pain
* Daily pain medication
* Frequent back pain
* On the job injury

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Miller, MD, Principal Investigator — Montefiore Medical Center; Benjamin W. Friedman, MD, MS, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CT-guided Intervention | Standard Medical Care
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — study terminated. no data collected. | 1 | 0

BASELINE CHARACTERISTICS:
Population: No data collected or analyzed because this study was terminated early due to low enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-guided Intervention | Standard Medical Care | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Impairment as Measured by the Roland Morris Disability Questionnaire
Description: The Roland Morris Disability Questionnaire (RMDQ) is a 24 item instrument that evaluates the impact of low back pain on one's daily life. It is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. Each question can be answered as either a "yes" or "no". The score ranges from 0 to 24 where a higher score reflects greater impairment and, therefore, worsening in the quality of life. The change in RMDQ is obtained by subtracting the RMDQ score at one week after discharge from the baseline score. The calculated mean and associated confidence interval values have been verified by staff statisticians.
Time Frame: Baseline and one week after emergency department discharge
Population: Study terminated due to low enrollment. No patient data was collected.
Arm/Group | CT-guided Intervention | Standard Medical Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Functional Disability Assessed Using Roland-Morris Scale
Description: The Roland Morris Disability Questionnaire (RMDQ) is a 24 item instrument that evaluates the impact of low back pain on one's daily life. It is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. Each question can be answered as either a "yes" or "no". The score ranges from 0 to 24 where a higher score reflects greater impairment and, therefore, increasing functional disability.
Time Frame: 1 month
Population: Study terminated due to low enrollment. No patient data was collected.
Arm/Group | CT-guided Intervention | Standard Medical Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Adverse Events
Description: Any adverse events since randomization. %s will be compared between groups
Time Frame: 1 week after discharge from emergency department
Population: Study terminated due to low enrollment. No patient data was collected.
Arm/Group | CT-guided Intervention | Standard Medical Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No data collected or analyzed because this study was terminated early due to low enrollment.
Arm/Group | CT-guided Intervention | Standard Medical Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes